CLINICAL TRIAL: NCT03797885
Title: An Observational Cross-sectional Study to Estimate the Prevalence of Cardiovascular Disease and CV Risk Factors in T2DM Patients Including a Retrospective Phase to Evaluate the Clinical Management of a Subgroup of Patients in the Hospital Setting in Portugal
Brief Title: A Study of People With Type 2 Diabetes Who Have Diseases That Affect the Heart and Blood Vessels. The Study Will Also Look at the Treatment of a Group of These People in Hospitals in Portugal
Acronym: PICT2RE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN2211-4435; U1111-1207-2878 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-01-02; First posted 2019-01-09 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with type 2 diabetes mellitus (T2DM): Patients with type 2 diabetes, at the hospital setting.
  Interventions: Other: No treatment given
- Patients with T2DM and established cardiovascular disease: Subgroup of patients with type 2 diabetes and established cardiovascular disease
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment is administered to the participants for this study

SUMMARY:
This study aims to estimate the number of patients with cardiovascular disease and risk factors in patients who had been diagnosed with type 2 diabetes mellitus. Simultaneously, this study also intends to obtain more information about the management of type 2 diabetes mellitus patients with established cardiovascular disease. This study is non-interventional, which means that will not require participant's further related visits or procedures. The study will collect the participant's clinical data from the current visit and, when applicable, within the last 3 years.

ELIGIBILITY:
Inclusion Criteria:

Main study population (Data collection - Prevalence):

* Signed Informed Consent Form (ICF) obtained before any study-related activities (study-related activities are any procedures related to recording of data according to protocol)
* Male or female patient, age greater or equal to 18 years at the time of signing ICF
* Patients diagnosed with type 2 diabetes

Subgroup (Data collection - Patient management):

* Patients followed at the hospital setting by the endocrinologist or internal medicine specialist (ambulatory diabetes management) and with available medical records, retrospectively within the last three years
* Patients with type 2 diabetes mellitus and established cardiovascular disease diagnosed at least three years ago

Exclusion Criteria:

* Previous participation in this study. Participation is defined as signed ICF
* Female patient who is pregnant or breast-feeding
* Patients with type 1 diabetes
* Participation in a clinical trial within the last 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 730 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Proportion of type 2 diabetes mellitus (T2DM) patients with cardiovascular risk factors (CVRFs) and/or established cardiovascular disease (CVD), regardless the date of diagnosis | Baseline (month 0)
  Proportion of subjects.
  CVRFs are defined as a history of one or more of the following criteria:
  * Overweight or obese
  * Family history of CVD (1st degree)
  * Hypertension
  * Hypercholesterolemia
  * Low high-density lipoproteins
  * Hypertriglyceridemia
  * Smoking habits
  * Sedentary lifestyle -as per Investigator discretion according to his/her normal practice.
  CVD is defined as a history of one or more of the following events:
  * Stroke
  * Transient ischaemic attack
  * Ischaemic heart disease including myocardial infarction
  * Congestive heart failure
  * Atrial fibrillation
  * Aortic aneurism
  * Peripheral or carotid artery disease

SECONDARY OUTCOMES:
Hypoglycaemic episodes | During 3 years before baseline (0 to -36 months)
  Number of episodes
Hyperglycaemic episodes | During 3 years before baseline (0 to -36 months)
  Number of episodes
Presence of T2DM complications (yes/no) | During 3 years before baseline (0 to -36 months)
  Number of patients for whom 'presence of T2DM complications' has been answered yes/no respectively
Types of T2DM complications | During 3 years before baseline (0 to -36 months)
  Types of T2DM complications: Retinopathy, Diabetic neuropathy (peripheral, autonomic), Diabetic nephropathy, Amputation.
Hospital appointments | During 3 years before baseline (0 to -36 months)
  Number of cardiology, ophthalmology, nephrology, and vascular surgery appointments
Hospitalisation episodes | During 3 years before baseline (0 to -36 months)
  Number of episodes
Emergency visits | During 3 years before baseline (0 to -36 months)
  Number of visits
Change in waist circumference | During 3 years before baseline (0 to -36 months)
  Measured in cm
Change in body mass index | During 3 years before baseline (0 to -36 months)
  Measured in kg/m^2
Change in blood pressure | During 3 years before baseline (0 to -36 months)
  Measured in mmHg
Change in urine albumin | During 3 years before baseline (0 to -36 months)
  Measured in mg/24 hours
Change in urine albumin | During 3 years before baseline (0 to -36 months)
  Measured in microgram/minute
Change in glycosylated hemoglobin (HbA1c) | During 3 years before baseline (0 to -36 months)
  Measured in mmol/mol
Change in HbA1c | During 3 years before baseline (0 to -36 months)
  Measured in %
Change in Estimated Glomerular Filtration Rate (eGFR) | During 3 years before baseline (0 to -36 months)
  Measured in mL/min/1.73 m^2
Change in total cholesterol | During 3 years before baseline (0 to -36 months)
  measured in mg/dl
Change in low-density lipoprotein cholesterol | During 3 years before baseline (0 to -36 months)
  measured in mg/dl
Change in high-density lipoprotein cholesterol | During 3 years before baseline (0 to -36 months)
  measured in mg/dl
Change in triglyceride | During 3 years before baseline (0 to -36 months)
  measured in mg/dl
Type of pharmacological treatment | During 3 years before baseline (0 to -36 months)
  Types of pharmacological treatment: Antidiabetics Antihypertensive Lipid lowering therapy Antiplatelet/anticoagulant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (11):
- Portugal (11):
  - Novo Nordisk Investigational Site, Almada
  - Novo Nordisk Investigational Site, Caldas da Rainha
  - Novo Nordisk Investigational Site, Leiria
  - Novo Nordisk Investigational Site, Lisbon
  - Novo Nordisk Investigational Site, Matosinhos Municipality
  - Novo Nordisk Investigational Site, Portimão
  - Novo Nordisk Investigational Site, Porto
  - Novo Nordisk Investigational Site, Viana do Castelo
  - Novo Nordisk Investigational Site, Vila Nova de Gaia
  - Novo Nordisk Investigational Site, Vila Real
  - Novo Nordisk Investigational Site, Viseu

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com